CLINICAL TRIAL: NCT06203379
Title: Effects of Preseason Neuromuscular Training Improves , Youth, Male Soccer Players
Brief Title: Efficacy of Neuromuscular Training in Youth Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-7993
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Exercise Training (Experimental)
  Interventions: Other: Neuromuscular Exercise Training
- Exercise Training (Active Comparator)
  Interventions: Other: control exercise

INTERVENTIONS:
Other: Neuromuscular Exercise Training — Neuromuscular Exercise Training
  Arms: Neuromuscular Exercise Training
Other: control exercise — Exercise Training
  Arms: Exercise Training

SUMMARY:
Soccer stands as one of the most widespread sports that ensures active participation . It has continued to grow and develop since its inception in all societies

DETAILED DESCRIPTION:
Footballers suffer injuries in various ways during training sessions and matches throughout the season due to excessive strain. Hence, numerous studies have investigated the injury sites and frequencies of footballers. According to these findings, it has been determined that young footballers experience more lower extremity injuries compared to professional footballers.

ELIGIBILITY:
Inclusion criteria:

* Being between the ages of 15-16
* Playing amateur football for at least 2 years
* Being a male athlete
* Voluntarily participate in the study
* Obtaining informed consent from them

Exclusion criteria:

* Bone fractures, fractures, ligament and muscle tears in the body.
* Has a systemic disease
* Having a serious injury in the last 3 months.
* Having any neurological problem

Ages: 15 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2024-01-14 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
vertical jump height | 8 weeks
  Optojump device was used for the assessment of jump height. Optojump is an optical sensor system used for sports and performance analysis. It accurately assesses athletes' fundamental parameters like jumping, speed, agility, and vertical leap to measure and enhance their physical abilities. The device uses a series of sensors and specialized software to monitor athletes' performance, enabling them to plan more effective training and continuously improve their performance.
jump duration (flight time) | 8 weeks
  Optojump device was used for the assessment of jump duration (flight time). Optojump is an optical sensor system used for sports and performance analysis. It accurately assesses athletes' fundamental parameters like jumping, speed, agility, and vertical leap to measure and enhance their physical abilities. The device uses a series of sensors and specialized software to monitor athletes' performance, enabling them to plan more effective training and continuously improve their performance.
Y Balance Test | 8 weeks
  The Y Balance Test evaluates an individual's dynamic balance, flexibility, and overall neuromuscular control. Commonly used in physiotherapy, sports medicine, and rehabilitation, it involves a series of movements where an individual maintains balance on one leg while reaching as far as possible with the other leg in various directions, forming a Y shape. Health professionals obtain valuable information about lower limb strength and stability by measuring the reached distances and assessing the ability to control multi-directional movements.
Fatigue Severity Scale | 8 weeks
  this scale comprises nine items. Participants rate their agreement with each statement on a scale from 1 to 7, where 1 indicates strong disagreement and 7 indicates strong agreement. A score of 4 or higher generally indicates severe fatigue
The Shuttle Run Test | 8 weeks
  It increases in difficulty as participants try to cover the specified distance within shorter intervals between shuttles. The number of completed shuttles reflects the individual's aerobic endurance level, serving as a common too for adjusting training programs and monitoring endurance levels for athletes and sports teams.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçehir University, Istanbul, Turkey (Türkiye)